CLINICAL TRIAL: NCT02764034
Title: Low Level Laser Therapy to Endometrial Cells: A Novel Approach to Increase Endometrial Proliferation and Enhance Endometrial Receptivity
Brief Title: Effect of Low Level Laser Therapy on Endometrial Cells: An In Vitro Study
Acronym: LLLT
Status: Available | Type: Expanded Access
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Abdelmageed El Faham, Doctor, National Research Centre, Egypt
Other Study IDs: effect of low level laser 001
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: Low level Laser; Tissue culture; Endometrial receptivity
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Device: Low level Laser diode machine — wavelength 635 Low level diode laser power control time control Continuous mode

SUMMARY:
The human endometrium is an extremely sensitive target. LLLT can enhance the proliferation rate of various cell lines, it produces higher rates of ATP, RNA, and DNA synthesis in stem cells and other cell lines. Thus, LLLT improves the proliferation of the cells without causing any cytotoxic effects.

The aim of this work is to assess the ability of low level laser therapy in enhancing endometrial proliferation and increasing endometrial receptivity.

A number of 120 human endometrial samples will be studied, and will be collected from 40 infertile women attending the infertility clinic at NRC. Each human endometrial sample will be divided into 3 plates, in order to establish 3 main groups of 40 culture plates for single laser exposure group versus 40 culture plates for multiple laser exposure group and 40 tissue culture plates for control samples, thus a total of 120 tissue culture plates will be studied, the study groups will be exposed to low level laser therapy and compared to their matched controls.. Assessment of number and size of cells after LLLT as a marker of normal proliferation and b) The expression of Integrin aVB3 "alpha v B3", MUC-1 and LIFand the development of pinopodes on the surface of epithelial cells as markers of endometrial receptivity and the detection of PTEN tumor suppressor gene as a marker of abnormal proliferation or premalignant condition will be performed to assess the effect of LLLT on the endometrial cell culture. This study might offer a new therapeutic modality which might increase endometrial thickness and enhance receptivity .

DETAILED DESCRIPTION:
Plan of work:

A number of 40 human endometrial samples will be collected from 40 infertile women attending the infertility clinic at the National Research Center (each sample will be divided into 3 culture plates; single exposure group, multiple exposure group and control group) and will be included in the study.

Each human endometrial sample will be divided into 3 plates, in order to establish 3 main groups of 40 culture plates for single laser exposure group versus 40 culture plates for multiple laser exposure group and 40 tissue culture plates for control samples, thus a total of 120 tissue culture plates will be studied, the study groups will be exposed to low level laser therapy and compared to their matched controls.

Timing of endometrial tissue sample:

Endometrial tissue biopsy will be performed in the early proliferative phase just after menstruation ceases (from day 5 to day8).

Consent A written informed consent will be obtained from each woman before the procedure. The consent will explain the purpose from the procedure, the aim from the research and the possible side effects.

Endometrial cell culture:

Endometrial biopsy strips will be collected from women included in the study. The endometrial biopsy strips will be taken from the uterine wall using pipelle.

Endometrial tissue will be transported to the laboratory in isolation media. Endometrial tissue will be stored at 4°C, and processed within 2-10 h.

Clusters of cells will be considered colonies when they become visible macroscopically and contain greater than 50 cells.

The same culture condition will be applied to both study and control samples. The tissue culture will be discarded after 14 days when the study will be completed.

Low level laser therapy will be wavelength 635nm diode laser, power of 40mw will be tested on cultured endometrial cells in Petri dish S.A. of 9.62cm2 with fluence rate of 4.2 J/cm2 in the continuous mode, depth of penetration at 635nm ranges from 1 to 6mm.

Tissue cultures in the study group will be divided into 2 groups; The 1st group will be composed of 40 tissue culture plates and will be exposed to the total fluence dose 4.2 J/cm2 in a single session of 16 minutes duration with low level therapy machine adjusted at power of 40mw. The 2nd group will be composed of another 40 tissue culture plates, they will be exposed to the same fluence rate but in multiple sessions ''3 sessions'', which will be performed every other day, each session will last for approximately 5.34 minutes using low level laser of power of 40mw to reach the same fluence dose of 4.2 J/cm2 after finishing the 3rd session.

Single versus multiple exposures of LLLT will be tested in the endometrial culture plates and will be compared to control group not exposed to laser. Comparison between single session exposure and multiple sessions' exposure is important in order to determine the benefits over the risk of multiple exposures sessions in thin endometrium in vivo, being an invasive procedure and requiring a fibro-optic probe insertion inside the uterus which might cause some discomfort to the patient and could be affected by patient's compliance.

RT-PCR Analysis technique and steps:

Real time PCR will be used to screen and detect the presence of endometrial implantation markers namely the expression of Integrin aVB3 "alpha v B3", MUC-1, LIF and also the expression of PTEN tumor suppressor gene as an early marker for premalignant endometrial disease.

Electron microscopy; Cells in tissue culture will be examined by electron microscope in order to detect the presence of pinopodes as a marker of increased endometrial receptivity.

ELIGIBILITY:
Inclusion Criteria:

Demographic:

* Women in child bearing period aging from 20 to 38 years.
* Only women up to 38 years will be included, to remove advanced age as a confounding factor that could affect the study results.
* BMI: > 20 and < 35 " BMI more 35 is excluded to remove any confounding factor related to increased BMI form the study"
* Human endometrial sample will be obtained from infertile women with the following conditions:

  * Recurrent IUI, IVF or ICSI Failure without any clear cause.
  * Women with unexplained infertility after exclusion of all other causes of infertility and exclusion of male factor.

Exclusion Criteria:

* Women with endometrial cancer or precancerous lesions.
* Women with any malignancy of the genital tract as vulval, vaginal, cervical, ovarian and other malignancies.
* Women undergoing dilatation and curettage due to the following conditions will be excluded:

  * Any pregnancy related pathology (eg, incomplete abortion, missed abortion, septic abortion, induced pregnancy termination, treatment and evaluation of gestational trophoblastic disease).
  * Dilatation and curettage for dysfunctional uterine bleeding; irregular bleeding or menorrhagia
  * Hormonal treatment or any medication that may affect the endometrium, including any patient received hormonal therapy in the 3 months preceding the study.
  * Before endometrial ablation for treatment of endometrial hyperplasia or perimenopausal bleeding.
* Tissues with proved precancerous or neoplastic changes in the endometrial sample will be discarded and eliminated before initiation of the study.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Amr H. El Noury, MD, FRCOG, Study Director — Cairo University; Marwa A. El Shaer, MD, Study Chair — Professor of Pathology at National Research Centre; Mona I. Morsy, MD, Study Director — Lecturer in Molecular Biology in National Institute of Laser and Enhanced Science; Osama M. Azmy, MD, FRCOG, Study Director — Professor of obstetrics and gynecology at National Research Centre
Locations (1):
- National Research Centre, Cairo, El Dokki, Egypt

REFERENCES:
- See also: 1. AlGhamdi KM, Kumar A, Moussa NA (2012). Low-level laser therapy: a useful technique for enhancing the proliferation of various cultured cells. Lasers Med Sci. Vol.27(1), pp.237-249. [PubMed] — http://PubMed
- See also: Barolet D (2008). Light-emitting diodes (LEDs) in dermatology. Semin Cutan Med Surg. Vol.27(4), pp.227-238. — http://PubMed
- See also: Avci P., Gupta A, Sadasivam M, Vecchio D., Pam Z, Pam N., and Hamblin M.R. (2013). Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg. Vol.32(1), pp.41-52 [PubMed] — http://PubMed
- See also: Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR (2012). The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. Vol.40 (2), pp.516-533. — http://PubMed